CLINICAL TRIAL: NCT05255757
Title: Social Network Interventions to Reduce Race Disparities in Living Kidney Donation
Brief Title: Network Interventions to Reduce Disparities in Living Kidney Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Pennsylvania (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan Daw, Associate Professor of Sociology and Demography, Penn State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 849197
Record Dates: First submitted 2021-10-10; First posted 2022-02-25 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: There are two interventions randomly assigned to participants in a factorial experimental design. The first intervention is the search intervention. In addition to the candidate survey, transplant candidates assigned to this intervention will be given information about the statistical likelihood that each member of their social network will be free of contraindications for living kidney donation. The second intervention is the script intervention, where in addition to the survey, transplant candidates will review a set of suggested talking points and an example script to guide discussion of potential living donation with members of their network. 25% of participants will be assigned to each of the following factorial experimental groups: no intervention, search intervention only, script intervention only, or both search and script intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No intervention (No Intervention): This group will only complete study survey and refer members of their family and social network for participation in a web survey.
- Script Intervention (Experimental): This group will complete the survey, refer members of their family and social network for participation in a web survey, and review a set of suggested talking points and an example script to guide discussion of potential living donation with members of their network.
  Interventions: Behavioral: Script Intervention
- Search Intervention (Experimental): This group will complete the candidate survey, refer members of their family and social network for participation in a web survey, and be given information about the statistical likelihood that each member of their social network will be free of contraindications for living kidney donation.
  Interventions: Behavioral: Search Intervention
- Both Search and Script Intervention (Experimental): This group will complete the candidate survey, refer members of their family and social network for participation in a web survey, be given information about the statistical likelihood that each member of their social network will be free of contraindications for living kidney donation, and review a set of suggested talking points and an example script to guide discussion of potential living donation with members of their network.
  Interventions: Behavioral: Script Intervention; Behavioral: Search Intervention

INTERVENTIONS:
Behavioral: Script Intervention — This intervention provides language to participants to allow them to discuss kidney transplantation with their social network.
  Arms: Both Search and Script Intervention; Script Intervention
Behavioral: Search Intervention — This group will complete the candidate survey, refer members of their family and social network for participation in a web survey, and be given information about the statistical likelihood that each member of their social network will be free of contraindications for living kidney donation.
  Arms: Both Search and Script Intervention; Search Intervention

SUMMARY:
For this current phase of the larger project, the investigators will survey transplant candidates as well as the participants family and friends to understand the barriers to volunteering and evaluation. This project will examine how network characteristics are associated with eventual living donor kidney transplant outcomes and test the efficacy of evidence-based interventions designed to assist kidney transplant candidates in participant donor search on a multi-center scale.

DETAILED DESCRIPTION:
The overall goal is to understand the process and assist participants who do not receive unsolicited offers to be evaluated as a living kidney donor in initiating and effectively conducting these critical conversations with participants kin and friends. In the search intervention, based on what they can tell investigators about the number, type, perceived health, perceived relationship, and potential willingness to donate, as well as analyses of data from the National Health and Nutrition Examination Survey (NHANES) investigators will counsel them on which members of participants family and friendship networks appear most biomedically promising as donors among the subset of these individuals that participants have not ruled out for known medical or perceived relationship reasons. In the rhetorical intervention, investigators will test non-coercive, promising verbal scripts that have proven promising in preliminary tests in vignette experiments in online and phone surveys.

AIM 1: Survey transplant candidates about their social network and transplant-related attitudes, knowledge, and characteristics; and randomize participants into one of two interventions or a control group.

AIM 2: Send network member participants a survey that measures potential donor attributes that are hypothesized to influence donation decisions, such as medical contraindications, blood type, health insurance status, and barriers to living donation.

AIM 3: Test whether participant social networks and interventions affect donation outcomes using medical records and follow-ups provided by Penn and UAB. Investigators will create the first predictive model of potential donor evaluation and actual donation. This information is critical to improve clinical practice and efforts to ethically influence the living donor search process.

ELIGIBILITY:
Inclusion Criteria:

* Are KT candidates at the University of Pennsylvania or University of Alabama-Birmingham OR were identified by KT candidate from the University of Pennsylvania or University of Alabama-Birmingham as a network member
* Are adults aged 18 or older
* Are able and willing to consent to participation in the survey

Exclusion Criteria:

* Person is not a KT candidate at University of Pennsylvania or University of Alabama-Birmingham OR was NOT identified by KT candidate from University of Pennsylvania or University of Alabama-Birmingham as a network member
* Individuals who are not yet 18
* Participant does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Received a living donor kidney transplant | up to 3 years
  Living donor kidney transplant received by patient
Received a deceased donor kidney transplant | up to 3 years
  Deceased donor kidney transplant received by patient
Death | up to 3 years
  Patient died during the follow-up period
Completed living kidney donor screening questionnaires | up to 3 years
  Number of completed living kidney donation screening questionnaires completed for patient
Preliminary approval from living kidney donor screening questionnaires | up to 3 years
  Number of completed living kidney donor screening that received preliminary approval for patient
Completed living kidney donor evaluations | up to 3 years
  Number of living kidney donor evaluations completed for patient
Approvals for living kidney donor candidacy | up to 3 years
  Number of completed living kidney donor evaluations that resulted in approved living kidney donor candidacy for patient

SECONDARY OUTCOMES:
Preference for living kidney donor | Immediate
  A set of survey questions asked both before and after the intervention, to assess intermediate attitude outcomes regarding preference for living kidney donor
Concerns about living kidney donation | Immediate
  A set of survey questions asked both before and after the intervention, to assess intermediate attitude outcomes regarding concerns for living kidney donation
Living donor kidney transplant willingness | Immediate
  A set of survey questions asked both before and after the intervention, to assess intermediate attitude outcomes regarding living donor kidney transplant willingness
Self-rated kidney transplant knowledge | Immediate
  Respondent is asked to rate their level of knowledge related to kidney transplantation.
Trust in medical institutions | Immediate
  Respondent is asked to rate their trust in medical institutions.
Religious views' effect on kidney transplant willingness | Immediate
  Respondent is asked how strongly they agree that their religious views affect their willingness to pursue a kidney transplant.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Penn Medicine-- University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No